CLINICAL TRIAL: NCT03330808
Title: Randomized Trials of Epidural Combined With General Anesthesia Versus General Anesthesia Alone to Evaluate the Changes of Blood Flow in Arterial Anastomosis of Free Flap Using Duplex Ultrasonography
Brief Title: Effect of Epidural Anesthesia on Blood Flow in Arterial Anastomosis of Free Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017-1200
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Free Tissue Flaps
MeSH Terms: interventions — Anesthesia, Epidural; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural with general anesthesia (Experimental): Epidural anesthesia with 0.2% ropivacaine 10 ml
  Interventions: Other: Epidural anesthesia
- General anesthesia alone (No Intervention): Sevoflurane and nitrous oxide.

INTERVENTIONS:
Other: Epidural anesthesia — After anesthesia induction, epidural catheter is inserted into lumbar epidural in epidural with general anesthesia group. A 10 ml of 0.2% ropivacaine should be given in epidural space via a catheter when anastomosis of free flap is finished in epidural with general anesthesia group.
  Other Names: Epidural anesthesia with ropivacaine
  Arms: Epidural with general anesthesia

SUMMARY:
Comparing the changes of arterial anastomotic blood flow between general anesthesia alone and general anesthesia with epidural anesthesia in patients who undergoing free flap transposition using Duplex ultrasound.

DETAILED DESCRIPTION:
Maintaining adequate blood flow is important on the success of free flap surgery. Epidural anesthesia can influence blood flow during surgery. Therefore, investigators aim to compare the effect of epidural anesthesia combined with general anesthesia and general anesthesia alone on blood flow in arterial anastomosis site of the free flap.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo free flap transfer under general anesthesia.
* 18 years of age or older, under 80 years of age
* Those who voluntarily agreed to participate in this clinical study

Exclusion Criteria:

* If the patient does not agree to participate in the study
* ASA physical status IV or higher
* If the patient was diagnosed with diabetes
* If the patient was diagnosed with chronic renal failure
* If the patient was diagnosed with peripheral vascular disease or hyperlipidemia
* If vasopressors or inotropics was used preoperatively.
* Contraindication of epidural anesthesia such as usage of anticoagulant or abnormalities of laboratory finding.
* If the researcher finds it to be inappropriate

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Maximal blood flow velocity | 30 minutes after flap arterial anastomosis
  Maximal blood flow velocity measured by using Duplex ultrasound

SECONDARY OUTCOMES:
Blood volume | 30 minutes after flap arterial anastomosis
  Blood volume measured by using Duplex ultrasound
Arterial blood pressure | 30 minutes after flap arterial anastomosis
  Arterial blood pressure measured monitors
Cardiac output | 30 minutes after flap arterial anastomosis
  Cardiac output measured monitors
Pulse pressure variability | 30 minutes after flap arterial anastomosis
  Pulse pressure variability measured monitors
Body temperature | 30 minutes after flap arterial anastomosis
  Body temperature measured monitors
Arterial carbon dioxide concentration | 30 minutes after flap arterial anastomosis
  Arterial carbon dioxide concentration measured arterial blood gas analysis
Free flap failure | Day 7 after free flap surgery
  Free flap failure after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wright CJ, Cousins MJ. Blood flow distribution in the human leg following epidural sympathetic blockade. Arch Surg. 1972 Aug;105(2):334-7. doi: 10.1001/archsurg.1972.04180080180030. No abstract available. PMID 5044554
- [Background] Tuman KJ, McCarthy RJ, March RJ, DeLaria GA, Patel RV, Ivankovich AD. Effects of epidural anesthesia and analgesia on coagulation and outcome after major vascular surgery. Anesth Analg. 1991 Dec;73(6):696-704. doi: 10.1213/00000539-199112000-00005. PMID 1952169
- [Background] Pallares LC, Deane CR, Baudouin SV, Evans TW. Strain gauge plethysmography and Doppler ultrasound in the measurement of limb blood flow. Eur J Clin Invest. 1994 Apr;24(4):279-86. doi: 10.1111/j.1365-2362.1994.tb01086.x. PMID 8050457
- [Background] Lou F, Sun Z, Huang N, Hu Z, Cao A, Shen Z, Shao Z, Yu P, Miao C, Wu J. Epidural Combined with General Anesthesia versus General Anesthesia Alone in Patients Undergoing Free Flap Breast Reconstruction. Plast Reconstr Surg. 2016 Mar;137(3):502e-509e. doi: 10.1097/01.prs.0000479933.75887.82. PMID 26910694
- [Background] Delis KT, Knaggs AL, Mason P, Macleod KG. Effects of epidural-and-general anesthesia combined versus general anesthesia alone on the venous hemodynamics of the lower limb. A randomized study. Thromb Haemost. 2004 Nov;92(5):1003-11. doi: 10.1160/TH04-04-0233. PMID 15543327